CLINICAL TRIAL: NCT04045405
Title: Phase I, Randomized, Double-blind, Placebo-controlled Study to Assess Safety, PK and PD Parameters of CDR132L in Patients With Stable Heart Failure of Ischemic Origin (NYHA 1- 3)
Brief Title: Clinical Study to Assess Safety, PK and PD Parameters of CDR132L
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardior Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR132L-FIH01; 2019-001291-10 (EudraCT Number)
Record Dates: First submitted 2019-07-23; First posted 2019-08-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDR132L (Experimental)
  Interventions: Drug: CDR132L
- Saline (Placebo Comparator)
  Interventions: Drug: CDR132L

INTERVENTIONS:
Drug: CDR132L — i.v. administration

SUMMARY:
This is a Phase I, randomized, double-blind, placebo-controlled study to assess safety, pharmacokinetics and pharmacodynamic parameters of CDR132L in patients with stable heart failure of ischemic origin (NYHA 1-3).

DETAILED DESCRIPTION:
Objectives:

Primary

• To assess the safety of one single and one repeated dose of CDR132L in patients with stable heart failure of ischemic origin (NYHA 1-3).

Secondary • To characterize the pharmacokinetic (PK) profile of CDR132L in patients with stable heart failure of ischemic origin.

Exploratory

• To determine the effect of CDR132L on pharmacodynamic (PD) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Stable heart failure of ischemic origin

Exclusion Criteria:

* Heart failure of non-ischemic origin (hypertensive heart disease, myocarditis, alcoholic cardiomyopathy and cardiac dysfunction due to rapid atrial fibrillation),

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [safety and tolerability] | 4 months
  The incidence and severity of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 4 months
  Pharmacokinetics parameter derived by non-compartmental methods to measure maximum observed plasma concentration (Cmax)
Time to reach maximum plasma concentration (Tmax) | 4 months
  Pharmacokinetics parameter derived by non-compartmental methods to measure time to maximum plasma concentration (Tmax)
Area under the curve (AUC0-t) | 4 months
  Pharmacokinetics parameter area under the plasma concentration-time curve from time zero to last detectable plasma concentration (AUC0-t)
Area under the curve (AUC0-inf) | 4 months
  Pharmacokinetics parameter area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf)
Blood clearance (CL) | 4 months
  Pharmacokinetics parameter to determin clearance considering terminal elimination rate
Half life (t1/2) | 4 months
  Pharmacokinetics parameter to determin half-life rate (t1/2)
Volume of distribution (Vdss) | 4 months
  Pharmacokinetics parameter

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Hauke, MD MFPM, Study Director — Cardior Pharmaceuticals GmbH CMO; Jorg Taubel, MD FFPM, Principal Investigator — Richmond Pharmacology Ltd CEO
Locations (1):
- Richmond Pharmacology Ltd., 1A Newcomen Street, London Bridge, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taubel J, Hauke W, Rump S, Viereck J, Batkai S, Poetzsch J, Rode L, Weigt H, Genschel C, Lorch U, Theek C, Levin AA, Bauersachs J, Solomon SD, Thum T. Novel antisense therapy targeting microRNA-132 in patients with heart failure: results of a first-in-human Phase 1b randomized, double-blind, placebo-controlled study. Eur Heart J. 2021 Jan 7;42(2):178-188. doi: 10.1093/eurheartj/ehaa898. PMID 33245749
- [Derived] Huang CK, Kafert-Kasting S, Thum T. Preclinical and Clinical Development of Noncoding RNA Therapeutics for Cardiovascular Disease. Circ Res. 2020 Feb 28;126(5):663-678. doi: 10.1161/CIRCRESAHA.119.315856. Epub 2020 Feb 27. PMID 32105576